CLINICAL TRIAL: NCT03895749
Title: A Double-Blind, Placebo-Controlled Parallel Study to Investigate the Effect of a Nitric Oxide Supplementation Product on Endothelial Dysfunction and Prehypertensive Adults
Brief Title: Effect of a Nitric Oxide Supplementation Product on Endothelial Dysfunction and Prehypertensive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hypertension Institute, Nashville (Other)
Collaborators: Neogenis Laboratories (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Neo40 ADMA
Record Dates: First submitted 2019-03-15; First posted 2019-03-29 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Phase II, randomized,double-blind, placebo-controlled 2 arm parallel
Who Masked: Participant, Care Provider, Investigator
Masking Description: placebo-controlled study material
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neo40 Daily (Active Comparator): Per Capsule: N5-carbamoylornithine 100 mg, crataegus laevigata 100 mg, L-ascorbic acid 50 mg, vitamin B-12 0.05 mg, vitamin C 50 mg.
  Interventions: Dietary Supplement: NEO40 Daily
- Placebo (Placebo Comparator): Per Capsule: Beet Juice concentrate, Carmine, Croscarmellose Sodium, D-Mannitol, Magnesium Stearate, Orange flavour, Silicon dioxide, Stevia rebaudiana leaf, Xylitol.
  Interventions: Dietary Supplement: NEO40 Daily

INTERVENTIONS:
Dietary Supplement: NEO40 Daily — Per Capsule: N5-carbamoylornithine 100 mg, crataegus laevigata 100 mg, L-ascorbic acid 50 mg, vitamin B-12 0.05 mg, vitamin C 50 mg.

SUMMARY:
The nitric oxide supplementation product, Neo40 Daily®, provides a dietary source of No2-. The product also allows for robust No2-reduction to NO from the extremely potent nitrite-reducing capacity of the polyphenols found in Hawthorne berry.(Bartsch et al., 1993) Neo40 Daily® is a unique product since it provides the dietary source of No2-, as well as the rate limiting No2- reduction activity.

DETAILED DESCRIPTION:
Neo40 Daily® facilitates both endothelial dependent and independent NO production. The acute effects of Neo40 Daily® have been demonstrated in hypertensive patients.(Zand et al., 2011) Within 30 minutes following a single dose of the Neo40 Daily®, a significant reduction in systolic/diastolic BP and vascular compliance was observed, as well as, 4 hours following treatment, a significant improvement in endothelial function was seen. Furthermore, it has been used in longer term clinical trials to show elevated plasma levels of No3• and No2·, indicating an increase in systemically available NO, and lower levels of triglycerides in an older population with cardiovascular risk factors.(Zand et al., 2011) This pilot study also demonstrated a trend towards reduced BP and improved quality of life among its prehypertensive participates (Biswas et al., 2015). This current clinical trial aims to expand on this pilot study and examine the effect of NO supplementation on a pre- and mildly hypertensive populations with endothelial dysfunction as measured by EndoPAr® and asymmetric dimethyl L-arginine (ADMA). In a double blinded placebo controlled parallel arm study, we will further investigate the effect of Neo40 Daily® on 40 pre- and mildly hypertensive subjects with regards to changes in blood pressure, endothelial dysfunction and other markers of NO availability and CVD risk.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with seated resting systolic blood pressures between 130-160 mmHg and diastolic between 85 and 100 mm Hg (inclusive) at screening visit
* Subjects with an elevated ADMA
* Agreement to maintain current level of physical activity and diet throughout the study
* Agrees to comply with study procedures including willingness to fast at least 12 hours before blood samples, abstain from alcohol two days prior to blood sampling and blood pressure measurement, abstain from coffee at least 14 hours before blood pressure

Exclusion Criteria:

* Females who are pregnant, breastfeeding or planning to become pregnant during the course of the study.
* Seated office systolic blood pressure ou side of the target range (systolic BP<130 mm Hg or >160 mmHg) or diastolic BP< 85 or 100 mm Hg at screening visit
* The use of natural health products for th treatment of hypertension within 2 weeks of screening
* Significant cardiac history defined as a h story of myocardial infarction (Ml); coronary angioplasty or bypass graft(s); Valvular isease or repair; unstable angina pectoris; transient ischemic attack (TIA); cerebrovascular accidents (CVA); congestive heart failure; or coronary artery disease (CAD)
* Type I diabetes
* Unstable medical conditions that in the opinion of the Principle Investigator preclude the subject from participating in the study
* Alcohol or drug abuse within the last 6 months
* Clinically significant abnormal laboratory results at screening
* Participation in a clinical research trial wi hin 30 days prior to randomization
* Allergy or sensitivity to study supplemen ingredients
* Individuals who are cognitively impaired nd/or who are unable to give informed consent
* Any other condition which in the lnvestig tor's opinion may adversely affect the subject's ability to complete the study or its meas res or which may pose significant risk to the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is the between-group changes from baseline (Day 0) to end of study (Day 30) in daytime mean systolic and diastolic BP. | 30 days
  The primary efficacy outcome to be analyzed is the between-group changes from baseline (Day 0) to end of study (Day 30) in daytime mean systolic and diastolic BP readings using AHA guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Houston, MD, Principal Investigator — Hypertension Institute
Locations (1):
- Hypertension Institute, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No